CLINICAL TRIAL: NCT05419713
Title: Visual Mechanisms of Intermediate Distance Space Perception During Self-motion
Brief Title: Intermediate Visual Space Perception
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, He Zijiang, Professor, University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 94.0302; R01EY033190 (NIH)
Record Dates: First submitted 2022-06-01; First posted 2022-06-15 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Vision

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Visual scences (Experimental): Lit target locations in visual environment will be varied and subjects' perceived locations will be measured.
  Interventions: Other: Visual Stimuli for Space Perception

INTERVENTIONS:
Other: Visual Stimuli for Space Perception — The visual environment (e.g., target locations and texture backgrounds) will be varied and human behavioral responses (judged distances) will be measured to reveal the space perception and cognitive processes underlying space perception and navigation.

SUMMARY:
The ability to judge the locations of various objects from oneself during self-motion in the intermediate distance range (~2-25m) is crucial for successful performance of activities of daily living, such as walking and driving. However, little is known about the mechanisms of visual space perception involved in judging distance, the focus of this project, in the planning and/or execution of self-motion in the natural 3D environment. The theoretical knowledge to be gained from this project will contribute to the scientific literature and provide insights into how eye and neurological defects could impair visual space perception, wayfinding, and mobility.

DETAILED DESCRIPTION:
Every day human subjects rely on their vision to judge the absolute distances of objects around them to plan and guide their actions, such as walking and driving. This, way-finding, process of ascertaining one's position and planning for possible routes of actions cannot be accomplished without reliable perception of visual space in the intermediate distance range (~2-25m from the observer). Thus, the broad long-term objective of this project is to uncover the mechanisms underlying intermediate distance space perception that supports distance judgment.

Yet, less is known about the underlying mechanisms of intermediate distance space perception compared to those of near space perception (<2m). Moreover, extant knowledge is predominantly obtained from testing static observers, making it difficult to generalize to the more common situation where observers plan and execute self-motion. The latter situation is more complex because self-motion is accompanied by retinal image motion of static objects in the surrounding environment, potentially requiring the visual system to simultaneously track the locations of all objects in the environment. The visual system also requires more processing capacity because it has to simultaneously compute the visual space representation, explore the environment, implement motor controls, etc. Clearly, both challenges - coding complexity and capacity limitation - could pose as potential threats to our ability to efficiently judge absolute distances and implement actions. This project hypothesizes the visual system overcomes both challenges by: (a) spatially updating the moving observer's position using an allocentric, world-centered spatial coordinate system for representing visual space, and (b) use spatial working memory (spatial-image) during spatial updating. The investigators will examine both hypotheses in three specific aims.

Aim 1: Investigate the implementation of the allocentric, world-centered spatial coordinate system

Aim 2: Investigate the factors affecting the spatial updating of visual space

Aim 3: Investigate the role of spatial-image memory in visual space perception

The psychophysical experiments will measure human behavioral responses in the real 3D environment. This approach allows for understanding of how humans' natural ecological niche, namely, the ground surface, both constrains and supports space perception and action in the real world. The investigators will test human observers' ability to judge target locations in impoverished visual environments under various conditions, such as while manipulating the observers' cognitive load (attention and memory), or available visual and idiothetic (vestibular and proprioception) information, while they plan and/or execute self-motion (walking). The outcomes of this research will advance the space perception literature, bridge theoretical knowledge of visual space perception and memory-directed navigation (cognitive maps), as well as reveal the influence of vestibular and somatosensory signals. In turn, the theoretical advancements provide insights for better understanding of intermediate distance space perception related to eye and visual impairments and their impacts on mobility in the real 3D environment.

ELIGIBILITY:
Inclusion Criteria:

* Adults (up to 40 years of age)
* Children (18 years and older)
* Normal, or corrected-to-normal, visual acuity (at least 20/20)
* Stereo acuity (<20 arc sec).

Exclusion Criteria:

* Self-reported history of visual and eye diseases
* Physical movement restrictions.
* Vulnerable populations such as pregnant women will be excluded owing to the extensive time commitment required of the subjects.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-09-30 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Visual mechanisms of intermediate distance space perception (distance) before and after self-motion | During procedure, an average of 10 sec.
  Subjects will judge perceived distances (cm) of test targets from themselves before self-motion to establish a baseline measure. Subjects will then undergo self-motion for an average of 10 sec, and stop at a predetermined location. Then subjects will again judge the perceived distance (cm) of test targets after the self-motion. The change in perceived distance (cm) from baseline will reveal if their perception is affected by environmental factors, internal perceptual process and/or cognitive process.
Visual mechanisms of intermediate distance space perception (height) before and after self-motion. | Druing procedure, an average of 10 sec.
  Subjects will judge perceived heights (cm) of test targets relative to the floor or ceiling before self-motion to establish a baseline measure. Subjects will then undergo self-motion for an average of 10 sec, and stop at a predetermined location. Then subjects will again judge the perceived height (cm) of test targets after the self-motion. The change in perceived height (cm) from baseline will reveal if their perception is affected by environmental factors, internal perceptual process and/or cognitive process.

CONTACTS AND LOCATIONS:
Overall Officials: Zijiang He, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States